CLINICAL TRIAL: NCT04068961
Title: New Strategies of Genetic Study of Patients With Oculocutaneous Albinism
Acronym: GENALB
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/31
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Oculocutaneous Albinism; Mutation
Keywords: CGH array chip; Homozygosity mapping
MeSH Terms: conditions — Albinism, Oculocutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples (2 blood tubes or 1 aliquot of DNA) are recorded in the DNA bank because were collected during the genetic consultation of these patients

INTERVENTIONS:
Other: Genetic analyzes — Analysis by CGH array, homozygotic cartography and candidate gene sequencing

SUMMARY:
The oculocutaneous albinism is an autosomal recessive condition associated with mutations in 4 genes. In 20% of patients no mutation is identified. The optimization of genetic analysis methods and the search for new genes involved will help improve the diagnosis in these patients.

DETAILED DESCRIPTION:
The oculocutaneous albinism is an autosomal recessive condition associated with mutations in 4 genes. In 20% of patients no mutation is identified. The optimization of genetic analysis methods and the search for new genes involved will help improve the diagnosis in these patients.

.

ELIGIBILITY:
Inclusion Criteria:

-Oculocutaneous albinism (diagnosis validated by a clinician at the initial genetic consultation and did not show mutations of the TYR, OCA2, TYRP1, SLC45A2 genes)

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having been examined during a genetic consultation, with Oculocutaneous Albinism
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2010-10-31 (Actual); Study Completion 2010-10-31 (Actual)

PRIMARY OUTCOMES:
Presence of a genetic anomaly | At the screening
  Analysis by CGH (Comparative Genomic Hybridization) array : The Log2 values of the patient / reference fluorescence intensity ratios (Log2R) are -1 in the case of a heterozygous deletion, 0.5 in the case of heterozygous duplication and 0 in the absence of rearrangement.
Identification of a genetic mutation | At the screening
  By sequencing candidate genes : homozygotic cartography and candidate gene sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Fanny MORICE-PICARD, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No